CLINICAL TRIAL: NCT01095263
Title: Assessment of Efficacy, Safety and Effects on Quality of Life of Deep Brain Stimulation to the Medial Forebrain Bundle in Patients With Treatment Resistant Major Depression (FORESEE: FOREbrain Stimulation dEprEssion)
Brief Title: Effects of Deep Brain Stimulation in Treatment Resistant Major Depression
Acronym: FORESEE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Thomas E. Schlaepfer, MD, Professor of Psychiatry and Psychotherapy, University Hospital, Bonn
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BSG-10-4711DBS
Record Dates: First submitted 2010-03-24; First posted 2010-03-30 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham then Stimulation (Experimental)
  Interventions: Device: DBS; Device: No Stimulation (Sham)
- Stimulation then Sham (Experimental)
  Interventions: Device: DBS; Device: No Stimulation (Sham)

INTERVENTIONS:
Device: DBS — 130Hz, 90us pulsewidth, 4V Amplitude
  Other Names: INS
Device: No Stimulation (Sham) — 130Hz, 90us pulsewidth, 0V Amplitude
  Other Names: INS

SUMMARY:
The investigators will investigate in a sham controlled design antidepressant effects and safety of DBS to the superolateral branch of the main medial forebrain bundle (slMFB).

DETAILED DESCRIPTION:
The target point for DBS in major depression disorder is located lateral to the ventral tegmental area (VTA) in the midbrain at the branching point of the superolateral branch (slMFB) from the main medial forebrain bundle (MFB).

The exact stimulation coordinates are:

MNI152 coordinates:

left: x(lat.)=-5, y(ap)=-14, z(vert.)=-8 right: x(lat.)=5, y(ap)=-14, z(vert.)=-9

MCP coordinates:

eft: x(lat.)=-6, y(ap)=-1, z(vert.)=-6 right: x(lat.)=4, y(ap)=-1, z(vert.)=-7

All coordinates refer to the MNI152 brain. Legend: slMFB = superolateral branch of medial forebrain bundle, MNI152=Montreal Neurologic Institute brain 152 coordinates, MCP = mid-commissural point coordinates, lat. = lateral, ap= antero-posterior, vert. = vertical.

More information can be found at: http://goo.gl/n9sWV

In addition to the described intervention, we will record EEG activity within the implanted regions during cognitive paradigms (Fell and Axmacher, Nat Rev Neurosci 2011). Specifically, we will investigate the neural mechanisms underlying classification learning, working memory and exploration of rewarded spatial locations and explore oscillatory responses following stimulation of the target regions. These experimental paradigms will be conducted on the first day after electrode implantation.

ELIGIBILITY:
Inclusion Criteria:

* Major depression (MD), severe, unipolar type
* German mother tongue
* Hamilton Depression Rating Scale (HDRS24) score of > 20
* Global Assessment of Function (GAF) score of < 45
* At least 4 episodes of MD or chronic episode > 2 years
* > 5 years after first episode of MD
* Failure to respond to

  * adequate trials (>5 weeks at the maximum recommended or tolerated dose) of primary antidepressants from at least 3 different classes;
  * adequate trials (>3 weeks at the usually recommended or maximum tolerated dose) of augmentation/combination of a primary antidepressant using at least 2 different augmenting/combination agents (lithium, T3, stimulants, neuroleptics, anticonvulsants, buspirone, or a second primary antidepressant);
  * an adequate trial of electroconvulsive therapy [ECT] (>6 bilateral treatments) and;
  * an adequate trial of individual psychotherapy (>20 sessions with an experienced psychotherapist).
* Able to give written informed consent
* No medical comorbidity
* Drug free or on stable drug regimen at least 6 weeks before study entry

Exclusion Criteria:

* Current or past nonaffective psychotic disorder
* Any current clinically significant neurological disorder or medical illness affecting brain function, other than motor tics or Gilles de la Tourette syndrome
* Any clinically significant abnormality on preoperative magnetic resonance imaging (MRI)
* Any surgical contraindications to undergoing DBS
* Current or unstably remitted substance abuse (aside from nicotine)
* Pregnancy and women of childbearing age not using effective contraception
* History of severe personality disorder

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Depression Severity assessed with Montgomery Asberg Depression Scale (MADRS) | 12 month after DBS stimulation onset
  Change in MADRS after 12 months as compared to mean baseline score. MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. It is used as an adjunct to the Hamilton Rating Scale for Depression (HAMD) and more sensitive to the changes in depression than the Hamilton Scale is.
  MADRS will be rated 3 times for baseline assessment, weekly during parameter optimization and monthly during follow-up. Reduction compared to baseline will be assessed after 12 months of DBS.

SECONDARY OUTCOMES:
Depression Severity rated with Hamilton Depression Rating Scale (HDRS24) | 12 month after DBS stimulation onset
  The Hamilton Rating Scale for Depression (HRSD), also known as the Hamilton Depression Rating Scale (HDRS) or abbreviated to HAM-D, is a multiple choice questionnaire that clinicians may use to rate the severity of a patient's major depression. The questionnaire rates the severity of symptoms observed in depression such as low mood, insomnia, agitation, anxiety and weight loss. The questionnaire is presently one of the most commonly used scales for rating depression in medical research.
  Measures will be taken at same time points as primary outcome measure.
Adverse Event Schedule | 12 month after DBS stimulation onset
  Adverse events will be recorded during the study using a structured questionnaire. All possible AEs are assessed in severity, duration and actions taken. 12 months after stimulation onset results will be compiled and rated as being due to the surgical procedure, device, or stimulation. SAEs will be discussed individually if a modification of study protocol is required.
Comprehensive neuropsychological test battery | 12 month after DBS stimulation onset

CONTACTS AND LOCATIONS:
Overall Officials: Volker Coenen, MD, Principal Investigator — University Hospital, Bonn; Thomas E. Schlaepfer, MD, Principal Investigator — University Hospital, Bonn
Locations (1):
- University Hospital Bonn, Bonn, Germany

REFERENCES:
- [Background] Coenen VA, Schlaepfer TE, Allert N, Madler B. Diffusion tensor imaging and neuromodulation: DTI as key technology for deep brain stimulation. Int Rev Neurobiol. 2012;107:207-34. doi: 10.1016/B978-0-12-404706-8.00011-5. PMID 23206684
- [Background] Coenen VA, Schlaepfer TE, Maedler B, Panksepp J. Cross-species affective functions of the medial forebrain bundle-implications for the treatment of affective pain and depression in humans. Neurosci Biobehav Rev. 2011 Oct;35(9):1971-81. doi: 10.1016/j.neubiorev.2010.12.009. Epub 2010 Dec 22. PMID 21184778
- [Result] Schlaepfer TE, Bewernick BH, Kayser S, Madler B, Coenen VA. Rapid effects of deep brain stimulation for treatment-resistant major depression. Biol Psychiatry. 2013 Jun 15;73(12):1204-12. doi: 10.1016/j.biopsych.2013.01.034. Epub 2013 Apr 3. PMID 23562618
- [Result] Coenen VA, Madler B, Schlaepfer TE. Reply to: medial forebrain bundle stimulation-speed access to an old or entry into a new depression neurocircuit? Biol Psychiatry. 2013 Dec 15;74(12):e45-6. doi: 10.1016/j.biopsych.2013.06.017. Epub 2013 Aug 2. No abstract available. PMID 23916389
- [Derived] Kilian HM, Meyer DM, Bewernick BH, Spanier S, Coenen VA, Schlaepfer TE. Discontinuation of Superolateral Medial Forebrain Bundle Deep Brain Stimulation for Treatment-Resistant Depression Leads to Critical Relapse. Biol Psychiatry. 2019 Mar 15;85(6):e23-e24. doi: 10.1016/j.biopsych.2018.07.025. Epub 2018 Sep 22. No abstract available. PMID 30253883
- See also: DBS target site description — http://tiny.cc/sl-mfb